CLINICAL TRIAL: NCT06810830
Title: A Randomized Controlled Trial on Internet-Based Cognitive Behavioral Therapy (iCBT) and Internet-Based Eye Movement Desensitization and Reprocessing Flash Technique (iEMDR-FT) for Improving Mental Health in Breast Cancer Patients
Brief Title: ICBT and IEMDR-FT for Mental Health in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Çiğdem Kınık, Principal Investigator, Psychologist PhD(c), Part time Lecturer, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180/2024; 180/2024 Ethics Approval (Other: Istanbul Okan University Ethics Committee)
Record Dates: First submitted 2025-01-04; First posted 2025-02-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Traumatic Stress; Anxiety; Quality of Lifte; Depression
Keywords: Breast cancer; internet-based cognitive behavioral therapy; EMDR; Flash Technique; psychological distress; quality of life
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model. Participants are randomly assigned to one of two interventions-an internet-based Cognitive Behavioral Therapy (iCBT) program or an internet-based EMDR Flash Technique (iEMDR-FT)-and both groups receive their respective treatments over the designated study period. Outcomes are assessed at baseline, post-intervention, and at a three-month follow-up. The trial is open-label (no masking), as both participants and researchers are aware of the assigned intervention. It is designed to compare the two arms directly to evaluate their differential effectiveness in reducing psychological distress among breast cancer patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iCBT Group (Experimental): Participants receive a 7-week internet-based Cognitive Behavioral Therapy (iCBT) program.
  Interventions: Behavioral: Internet-Based Cognitive Behavioral Therapy (iCBT)
- iEMDR-FT Group (Experimental): Participants receive a 3-session internet-based EMDR Flash Technique (iEMDR-FT) within a one week.
  Interventions: Behavioral: Internet-Based EMDR Flash Technique (iEMDR-FT)

INTERVENTIONS:
Behavioral: Internet-Based Cognitive Behavioral Therapy (iCBT) — A structured 7-week program focusing on cognitive restructuring, stress management, and emotional regulation.
  Arms: iCBT Group
Behavioral: Internet-Based EMDR Flash Technique (iEMDR-FT) — A 3-session protocol adapted to minimize re-exposure to distressing cancer-related memories through rapid bilateral stimulation and positive imagery.
  Arms: iEMDR-FT Group

SUMMARY:
This study aims to compare the effectiveness of two internet-based therapy approaches in improving psychological well-being and reducing distress among patients diagnosed with breast cancer. Participants will be randomly assigned to one of two groups: a 7-week internet-based Cognitive Behavioral Therapy (iCBT) program or a 3-session internet-based Eye Movement Desensitization and Reprocessing Flash Technique (iEMDR-FT) within a week. Both interventions will be delivered online in a group format under the guidance of experienced therapists.

Participants' mental health status-including anxiety, depression, traumatic stress, fear of cancer recurrence, and overall quality of life-will be assessed before the intervention, immediately after completion, and again at a 3-month follow-up. The results of this study are expected to provide valuable insights into how digital psychotherapy methods can help breast cancer patients cope with emotional challenges during their treatment. The findings will also inform the development of future online psychosocial support models in oncology.

DETAILED DESCRIPTION:
Breast cancer is widely considered a complex condition that entails profound psychological repercussions alongside physical challenges. In addition to the stress of undergoing medical treatments, many patients develop an intense fear of cancer recurrence (FCR), depressive and anxious states, and symptoms that may meet the criteria for posttraumatic stress disorder (PTSD). Given these extensive emotional burdens, structured psychological interventions have emerged as vital components of comprehensive oncological care. While Cognitive Behavioral Therapy (CBT) is established as the gold standard for reducing anxiety and depression, emerging trauma-focused therapies-such as Eye Movement Desensitization and Reprocessing (EMDR)-are increasingly recognized for their efficacy in addressing cancer-related traumatic stress.

Among EMDR-based interventions, the Flash Technique (FT) represents an innovative adaptation designed to minimize the discomfort of processing traumatic memories. Unlike traditional EMDR protocols, which may require individuals to recall and discuss disturbing events in detail, the Flash Technique uses brief exposures to distressing imagery, followed by rapid bilateral stimulation and positive recall. These "flashes" can quickly desensitize the emotional intensity of cancer-related memories while reducing the risk of re-traumatization. Early studies on the Flash Technique have shown promise in alleviating traumatic symptoms in non-cancer populations, highlighting the method's potential to offer quick, effective relief from emotionally charged recollections. However, there is a notable lack of research exploring its efficacy specifically in patients with breast cancer.

This randomized controlled trial (RCT) is the first known study to directly compare the Flash Technique, adapted for online delivery (iEMDR-FT), with an internet-based CBT program (iCBT) in breast cancer patients. Participants are randomly assigned to one of two groups: a 7-week iCBT program or a 3-session iEMDR-FT protocol. The iCBT program focuses on cognitive restructuring, stress management, and emotional regulation skills tailored to address the unique challenges of cancer-related thought patterns (e.g., catastrophic thinking, fear of recurrence). In contrast, the iEMDR-FT group engages in low-intensity trauma processing, wherein participants briefly recall cancer-related distressing scenes, then undergo sets of rapid bilateral stimulation combined with positive imagery ("flash" sets). This approach aims to swiftly reduce traumatic arousal without requiring the prolonged confrontation of painful memories often associated with traditional trauma therapies.

Both interventions are delivered online in a group format, guided by experienced therapists. Assessments include measures of posttraumatic stress (PCL-5), fear of cancer recurrence, depression-anxiety-stress (DASS-21), and quality of life (WHOQOL-BREF). Data are collected at baseline, immediately post-intervention, and three months post-intervention to evaluate both immediate and sustained changes in participants' mental health status. By comparing these two distinct therapeutic modalities, the study seeks to determine whether the rapid, minimal-exposure Flash Technique offers advantages over-or is equivalent to-the more extended, structured cognitive framework of CBT.

The outcomes of this investigation may fill a critical gap in the current literature by clarifying the practical utility, safety, and acceptability of online EMDR Flash Technique in an oncology setting. If iEMDR-FT proves to be equally effective or superior to iCBT in reducing traumatic stress, fear of cancer recurrence, and emotional distress, it could represent a valuable, time-efficient option for treating psychological sequelae in breast cancer. Conversely, if iCBT demonstrates better long-term gains in certain domains-such as cognitive restructuring of illness-related beliefs-this will inform clinicians about the relative strengths of each intervention. Ultimately, this study is poised to provide evidence-based guidance for mental health professionals and oncology teams in selecting or integrating internet-based interventions, thereby contributing to more flexible and patient-centered psychosocial care for individuals coping with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Age: 18 to 65 years. Diagnosis: Diagnosed with breast cancer (any stage as determined by the treating oncologist, or specify Stage I-III, etc.).

Medical Status: Currently under medical follow-up for breast cancer or in remission (as appropriate for the study's design).

Language Proficiency: Able to read and write in Turkish (or the language used for the intervention materials).

Technical Requirements: Has stable internet access and is willing to participate in online group sessions.

Consent: Provides informed consent to participate in the study.

Exclusion Criteria:

Severe Psychiatric Disorders: Presence of a severe psychiatric disorder (e.g., active psychosis, bipolar disorder in a severe manic phase) that would impede participation in psychotherapy.

Neurological or Cognitive Impairment: Any significant neurological impairment or cognitive dysfunction that interferes with comprehension of online materials.

Confounding Study Participation: Concurrent enrollment in another clinical trial involving psychological or behavioral interventions that might confound study outcomes.

Attendance Issues: Inability or unwillingness to attend scheduled online group sessions.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change in PTSD Symptom Severity (PCL-5) | Baseline (Pre-Intervention), Post-Intervention (iCBT: Week 7; iEMDR-FT: after 3 sessions in one week, measured one week after the final session), and 3 Months Post-Intervention.
  PTSD symptom severity was assessed using the Posttraumatic Stress Disorder Checklist-5 (PCL-5), developed based on DSM-5 diagnostic criteria. The PCL-5 total score ranges from 0 to 80; a higher score reflects more severe posttraumatic stress symptoms. The change in score between pre-intervention, post-intervention, and the 3-month follow-up measurements indicates improvement in posttraumatic stress symptoms among participants in the two different internet-based therapy groups (iCBT and iEMDR-FT).

SECONDARY OUTCOMES:
Change in Depression, Anxiety, and Stress Levels (DASS-21) | Baseline (Pre-Intervention), Post-Intervention (within one week), 3-Month Follow-Up.
  Description: The Depression Anxiety Stress Scales-21 (DASS-21) is a 21-item self-report tool that measures levels of depression, anxiety, and stress. Each subscale contains seven items scored on a 4-point Likert scale (0-3). Higher scores indicate greater symptom severity. Assessments will be conducted at Baseline (Pre-Intervention), Post-Intervention (within one week), and 3 Months Post-Intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After the publication of the primary results, de-identified individual participant data will be made available upon request to qualified researchers via an institutional data-sharing agreement. Data will be accessible for analyses related to the aims of this study and subject to ethical approval. Requests can be submitted to the Principal Investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Start date: Immediately after publication of primary study results End date: Data will be available for 5 years following publication, after which archiving or removal from the repository may occur.
Access Criteria: Qualified researchers should contact the Principal Investigator at psk.cigdem@gmail.com to request access. A data use agreement must be signed to ensure compliance with privacy regulations and ethical guidelines.

REFERENCES:
- See also: An RCT found iEMDR-FT effectively reducing traffic-accident trauma, depression, anxiety, stress, and boosting quality of life with brief "flash" exposures and minimal emotional confrontation. — https://pubmed.ncbi.nlm.nih.gov/35401305/